CLINICAL TRIAL: NCT06021990
Title: Role of Clopidogrel in Preventing Exacerbations in Patients With Severe COPD: An Open-label Randomized Controlled Trial.
Brief Title: Clopidogrel for the Prevention of Exacerbations in Severe COPD
Acronym: CLOPEX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Collaborators: Pakistan Chest Society, Pakistan (Unknown)
Responsible Party: Principal Investigator, Muhammad Imran, Assistant Professor, Lady Reading Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 804/LRH/MTI
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: COPD; COPD Exacerbation Acute
Keywords: COPD; Acute exacerbation; Clopidogrel; Randomised Clinical Trial; prevention; CLOPEX; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Clopidogrel

STUDY DESIGN:
Intervention Model Description: After assessing eligibility and consent patients will be randomly assigned to either the intervention arm or control arm. The control arm would be standard of care treatment according to GOLD guidelines and approved by the Pakistan Chest Society. The intervention arm will take Clopidogrel 75mg dail according the study prototcol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clopidogrel group (Experimental): The clopidogrel group will receive the intervention under study (clopidogrel 75mg once daily post-meal) for the study period along with the standard of care treatment as approved by the hospital based on national and international guidelines.
  Interventions: Drug: Clopidogrel Bisulfate 75Mg Tab
- Standard of Care (No Intervention): The standard of care will receive treatment as approved by the hospital based on national and international guidelines.

INTERVENTIONS:
Drug: Clopidogrel Bisulfate 75Mg Tab — Severe COPD patients who meet eligibility criteria will be given Clopidogrel Bisulfate 75 mg Tablet daily, along with standard of care treatment till the completion of the study duration or any side effects that warrants stoppage of the drug
  Other Names: clopidogrel; Plavix
  Arms: Clopidogrel group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a debilitating respiratory disorder characterized by gradual and progressive airflow limitation. It has been hypothesized that clopidogrel may have a role in reducing the exacerbation of COPD by reducing thromboembolic events. Several observational studies have found that taking clopidogrel reduces the likelihood of COPD exacerbations in patients with the disease. The study being conducted will be a randomized control trial, from March 2023 to March 2024 in the department of pulmonology, LRH. The aim of the study is to determine the role of clopidogrel in reducing the frequency of exacerbation in COPD patients compared to controls. The sampling will be done by non-probability consecutive sampling and the patients will be randomly allocated in study and control groups. Both the groups will be followed at the 3rd, 6th, and 12th months of the treatment and will be compared for the outcomes.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a debilitating respiratory disorder characterized by gradual and progressive airflow limitation. It is a huge worldwide health issue as well as a major cause of morbidity and mortality. Currently, it is the third leading cause of death. Exacerbations, or abrupt worsening of symptoms that necessitate medical treatment, are common in people with severe COPD. Exacerbations negatively influence patients' quality of life and are linked to higher healthcare utilization and mortality.

Clopidogrel is a widely used antiplatelet medication that works by inhibiting platelet aggregation by blocking the P2Y12 receptor. Clopidogrel's potential benefits in the treatment of COPD have piqued the curiosity of researchers in recent years. According to the hypothesis, Clopidogrel may lower the incidence of exacerbations by reducing thromboembolic events, which are prevalent causes of exacerbations in COPD.

Several observational studies have found that taking clopidogrel reduces the likelihood of COPD exacerbations in patients with the disease. A meta-analysis on the reduction of all-cause mortality in COPD patients concluded that mortality might be significantly lower in COPD patients receiving antiplatelet treatment. However, because of confounding considerations, the findings of these observational studies should be regarded with caution. To confirm the potential benefits of clopidogrel in lowering COPD exacerbations, randomized controlled studies (RCTs) are required. Only a few RCTs have been undertaken to date, with inconsistent outcomes.

The inconsistent findings of the RCTs show the need for additional studies to determine the role of clopidogrel in reducing COPD exacerbations. Larger, well-designed RCTs are required to offer more firm information on the possible benefits and dangers of clopidogrel in this patient population. The RCTs should also consider clopidogrel's potential side effects, such as bleeding, which may be especially concerning in COPD patients who are frequently on numerous drugs and may have comorbidities such as cardiovascular disease.

Finally, the role of clopidogrel in lowering exacerbations in patients with severe COPD remains unknown. Observational studies suggest that clopidogrel may have some benefits, while RCT results are mixed. More research is needed to determine clopidogrel's safety and efficacy in this patient population.

The results of the study if successful, will have two impacts. First, it will help reduce the financial burden on our healthcare system. Second, it will improve patients' quality of life by less frequent hospital visits with lowered mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe COPD (GOLD stage III or IV based on FEV1)
* Patients with a history of at least one exacerbation in the past year.
* Patients who are able to understand and provide informed consent.
* Patients willing and able to comply with the study protocol and attend follow-up visits.
* Patients who are between the ages of 40 and 80 years.
* Either gender

Exclusion Criteria:

* Patients who have previously experienced serious medical issues, like a recent heart attack or stroke (within six months),
* Patients who are known to be hypersensitive to clopidogrel.
* People who have a history of gastrointestinal bleeding or any other health issue that could make them more likely to bleed.
* Women who are pregnant or nursing.
* Patients who are being treated with additional antiplatelet or anticoagulant medications.
* Patients who are being treated with clopidogrel for any other indication.
* People who suffer from severe renal or liver illness.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of acute exacerbations of COPD | 28 days
  The rate of COPD exacerbations during a 12-month period, which is characterised as a worsening of symptoms for less than 14 days needing systemic corticosteroids and/or antibiotics as treatment or admission to hospital for the symptoms, will be the main outcome indicator.

SECONDARY OUTCOMES:
The number of hospitalisations for COPD-related exacerbations | 28 days
  The number of hospitalizations required for acute exacerbation of COPD will be compared in both the intervention arm and control arm.
Change in forced expiratory volume in one second (FEV1) | 28 days
  The changes in FEV1 measured with a spirometer during the follow-up visits will be compared between the intervantion arm and the control arm till the completion of the study
Death | 12 months
  Mortality and survival will be compared between the intervention arm and the control arm till the completion of the study
Quality of life as measured by the St. George's Respiratory Questionnaire (SGRQ) | 28 days
  Quality of life as measured by the St. George's Respiratory Questionnaire (SGRQ) will be compared between the intervention arm and the control arm till the completion of the study. Calculated results include four scores: symptoms, activity, impacts, and total. Better health is indicated by lower scores. Maximum raw scores are as follows: 662.5, 1209.1, 2117.8, and 3989.4

CONTACTS AND LOCATIONS:
Overall Officials: Zafar Iqbal, MBBS, MCPS, FCPS, DHPE, Study Chair — Lady Reading Hospital, Pakistan
Locations (2):
- Pakistan (2):
  - Pulmonology Department, Lady Reading Hospital, Peshawar, Peshawar, Khyber Pakhtunkhwa
  - Saidu Teaching Hospital, Swat, Swāt, Khyber Pakhtunkhwa

REFERENCES:
- [Background] Pahal P, Hashmi MF, Sharma S. Chronic Obstructive Pulmonary Disease Compensatory Measures. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK525962/ PMID 30247837
- [Background] Murarescu ED, Mitrofan EC, Mihailovici MS. Chronic obstructive pulmonary disease in a new concept. Rom J Morphol Embryol. 2007;48(3):207-14. PMID 17914487
- [Background] Kim V, Aaron SD. What is a COPD exacerbation? Current definitions, pitfalls, challenges and opportunities for improvement. Eur Respir J. 2018 Nov 15;52(5):1801261. doi: 10.1183/13993003.01261-2018. Print 2018 Nov. PMID 30237306
- [Background] Beekman E, Mesters I, Hendriks EJ, Muris JW, Wesseling G, Evers SM, Asijee GM, Fastenau A, Hoffenkamp HN, Gosselink R, van Schayck OC, de Bie RA. Exacerbations in patients with chronic obstructive pulmonary disease receiving physical therapy: a cohort-nested randomised controlled trial. BMC Pulm Med. 2014 Apr 26;14:71. doi: 10.1186/1471-2466-14-71. PMID 24767519
- [Background] Damman P, Woudstra P, Kuijt WJ, de Winter RJ, James SK. P2Y12 platelet inhibition in clinical practice. J Thromb Thrombolysis. 2012 Feb;33(2):143-53. doi: 10.1007/s11239-011-0667-5. PMID 22183178
- [Background] Kunadian V, Chan D, Ali H, Wilkinson N, Howe N, McColl E, Thornton J, von Wilamowitz-Moellendorff A, Holstein EM, Burns G, Fisher A, Stocken D, De Soyza A; APPLE COPD-ICON2 Trial Investigators. Antiplatelet therapy in the primary prevention of cardiovascular disease in patients with chronic obstructive pulmonary disease: protocol of a randomised controlled proof-of-concept trial (APPLE COPD-ICON 2). BMJ Open. 2018 May 26;8(5):e020713. doi: 10.1136/bmjopen-2017-020713. PMID 29804061
- [Background] Pavasini R, Biscaglia S, d'Ascenzo F, Del Franco A, Contoli M, Zaraket F, Guerra F, Ferrari R, Campo G. Antiplatelet Treatment Reduces All-Cause Mortality in COPD Patients: A Systematic Review and Meta-Analysis. COPD. 2016 Aug;13(4):509-14. doi: 10.3109/15412555.2015.1099620. Epub 2015 Dec 17. PMID 26678708